CLINICAL TRIAL: NCT05320380
Title: A PedAL/EuPAL Phase 1/2 Trial of IMGN632 in Pediatric Patients With Relapsed or Refractory Leukemia
Brief Title: A Study of the Drug IMGN632 in Children With Leukemia That Has Come Back After Treatment or is Difficult to Treat
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn per CS0150757
Sponsor: Children's Oncology Group (Network)
Collaborators: ImmunoGen, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APAL2020B; NCI-2022-02157 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); APAL2020B (Other: Children's Oncology Group); APAL2020B (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Acute Myeloid Leukemia; Recurrent B Acute Lymphoblastic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Recurrent T Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory Mixed Phenotype Acute Leukemia; Refractory T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Biopsy; Cytarabine; fludarabine phosphate; Hydrocortisone; hydrocortisone hemisuccinate; CPX-351; Injections; Daunorubicin; Liposomes; Methotrexate; merphos; Prednisolone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Phase I non-randomized study followed by a phase II randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (IMGN632) (Experimental): Patients receive IMGN632 IV on days 1 and 22. Treatment repeats every 42 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-CD123 ADC IMGN632
- Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine) (Experimental): CYCLE 1: Patients receive IMGN632 IV on days 1 and 22 and CPX-351 IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients with CNS1 also receive ITT consisting of methotrexate IT, hydrocortisone or prednisolone IT, and cytarabine IT on day 0 of cycle 1 (NOTE: Patients who received IT cytarabine or ITT at time of diagnostic LP do not need to repeat ITT on day 0 if given within 7 days of starting protocol therapy). Patients with CNS2 receive ITT QW until the CSF is clear for a maximum of 6 ITT treatments in the absence of disease progression or unacceptable toxicity.
  CYCLE 2: Patients receive ITT on day 0, IMGN632 IV on days 1 and 22, fludarabine IV over 30 minutes QD on days 1-5, and cytarabine IV over 1-3 hours QD on days 1-5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-CD123 ADC IMGN632; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Drug: Fludarabine Phosphate; Drug: Hydrocortisone Sodium Succinate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Drug: Methotrexate; Drug: Prednisolone
- Cohort 3, Arm A (CPX-351, fludarabine, cytarabine) (Active Comparator): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 of cycle 1 in the absence of disease progression or unacceptable toxicity. Patients then receive fludarabine IV over 30 minutes QD on days 1-5 of cycle 2 and cytarabine IV over 1-3 hours QD on days 1-5 of cycle 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Fludarabine Phosphate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine
- Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632) (Experimental): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 of cycle 1 and IMGN632 IV on days 1 and 22 of cycle 1 in the absence of disease progression or unacceptable toxicity. Patients then receive fludarabine IV over 30 minutes QD on days 1-5 of cycle 2, cytarabine IV over 1-3 hours QD on days 1-5 of cycle 2, and IMGN632 IV on days 1 and 22 of cycle 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-CD123 ADC IMGN632; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Cytarabine; Drug: Fludarabine Phosphate; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Anti-CD123 ADC IMGN632 — Given IV
  Arms: Cohort 1 (IMGN632); Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine); Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration/biopsy
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine); Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632)
Drug: Cytarabine — Given IT and IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine); Cohort 3, Arm A (CPX-351, fludarabine, cytarabine); Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine); Cohort 3, Arm A (CPX-351, fludarabine, cytarabine); Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632)
Drug: Hydrocortisone Sodium Succinate — Given IT
  Other Names: (11beta)-21-(3-Carboxy-1-oxopropyl)-11,17-dihydroxypregn-4-ene-3,20-dione, Monosodium Salt; A-Hydrocort; Buccalsone; Corlan; Cortisol Sodium Succinate; Cortop; Efcortelan; Emergent-EZ; Flebocortid; Hidroc Clora; Hycorace; Hydro-Adreson; Hydrocort; Hydrocortisone 21-Sodium Succinate; Hydrocortisone Na Succinate; Kinogen; Nordicort; Nositrol; Sinsurrene; Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine)
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine); Cohort 3, Arm A (CPX-351, fludarabine, cytarabine); Cohort 3, Arm B (CPX-351, fludarabine, cytarabine, IMGN632)
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine)
Drug: Prednisolone — Given IT
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
  Arms: Cohort 2 (IMGN632, CPX-351, ITT, fludarabine, cytarabine)

SUMMARY:
This phase I/II trial finds the highest safe dose of IMGN632 that can be given with other chemotherapy without causing severe side effects, studies what kind of side effects IMGN632 may cause, and determines whether IMGN632 is a beneficial treatment for leukemia in children that has come back after treatment or is difficult to treat. IMGN632 is a monoclonal antibody linked to a chemotherapy drug. IMGN632 is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD123 receptors, and delivers the chemotherapy drug to kill them. Giving IMGN632 with other chemotherapy may cause the leukemia to stop growing or to shrink for a period of time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of anti-CD123 ADC IMGN632 (IMGN632) monotherapy in pediatric patients with second or greater relapse of CD123 positive leukemia or CD123 positive leukemia refractory to relapse therapy. (Cohort 1 [Monotherapy Phase 1]) II. To assess the flow-based overall response rate (complete remission [CR]/CR with incomplete blood count recovery [CRi]/CR with partial recovery of platelet count [CRp]) in patients with acute myeloid leukemia (AML) treated with IMGN632. (Cohort 1 [Monotherapy Phase 1]) III. To determine the safety, feasibility, and RP2D of IMGN632 in combination with liposome-encapsulated daunorubicin-cytarabine (DAUNOrubicin and cytarabine liposome) in pediatric patients with first relapse of CD123 positive AML. (Cohort 2 [Combination Therapy Dose Finding]) IV. To compare the minimal residual disease (MRD) negative flow-based overall response rate (CR/CRi/CRp) in pediatric patients with first relapse of CD123 positive AML randomized to two cycles of therapy including DAUNOrubicin and cytarabine liposome followed by fludarabine phosphate (fludarabine)/cytarabine with or without IMGN632. (Cohort 3 [Randomized Phase 2])

SECONDARY OBJECTIVE:

I. To characterize the pharmacokinetics of IMGN632 in a pediatric population. (Cohort 1 [Monotherapy Phase 1])

EXPLORATORY OBJECTIVES:

I. To describe the anti-leukemic activity (morphologic and flow-based CR/CRp/CRi after up to two cycles, rates of MRD negative response after up to 2 cycles, event free survival [EFS] and overall survival [OS]) of IMGN632 in patients with multiply relapsed or refractory relapsed pediatric leukemia including AML, B-cell acute lymphoblastic leukemia [ALL], T-cell ALL and mixed phenotype acute leukemia (MPAL). (Cohort 1) II. To describe the EFS, OS, cumulative incidence of relapse, and rate of subsequent stem cell transplant for patients with first relapse of AML randomized to treatment with up to two cycles of chemotherapy with or without IMGN632. (Cohort 3) III. To determine if CD123 expression on leukemic blasts (assessed by flow cytometry) correlates with clinical response to IMGN632. (All Cohorts) IV. To determine the cumulative incidence of left ventricular systolic dysfunction (LVSD), defined as an absolute decline in EF by >= 10% to an ejection fraction (EF) value of < 50%, or an absolute decline in shortening fraction (SF) by >= 4% to an SF value of < 25%, within 1 year of initiation of DAUNOrubicin and cytarabine liposome based therapy for relapsed pediatric AML.

V. To describe safety (adverse events) in pediatric leukemia patients treated with IMGN632 including long-term safety events related to treatment for up to 5 years. (All Cohorts)

OUTLINE: This is a phase I, dose-escalation study of IMGN632 followed by a phase II study. In phase I, patients with second or greater relapse or refractory relapsed disease of AML, B-ALL, T-ALL or MPAL with CD123 expression are assigned to Cohort I, while patients with CD123 positive AML in first relapse are assigned to Cohort II. In phase II, patients with first relapse of CD123 positive AML are assigned to Cohort III.

COHORT 1: Patients receive IMGN632 intravenously (IV) on days 1 and 22. Treatment repeats every 42 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

COHORT 2:

CYCLE 1: Patients receive IMGN632 IV on days 1 and 22 and liposome-encapsulated daunorubicin-cytarabine (CPX-351) IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. Patients with CNS1 also receive intrathecal triple therapy (ITT) consisting of methotrexate intrathecally (IT), hydrocortisone or prednisolone IT, and cytarabine IT on day 0 of cycle 1 (NOTE: Patients who received IT cytarabine or ITT at time of diagnostic lumbar puncture [LP] do not need to repeat ITT on day 0 if given within 7 days of starting protocol therapy). Patients with CNS2 receive ITT once weekly (QW) until the cerebrospinal fluid (CSF) is clear for a maximum of 6 ITT treatments in the absence of disease progression or unacceptable toxicity.

CYCLE 2: Patients receive ITT on day 0, IMGN632 IV on days 1 and 22, fludarabine IV over 30 minutes once daily (QD) on days 1-5, and cytarabine IV over 1-3 hours QD on days 1-5 in the absence of disease progression or unacceptable toxicity.

COHORT 3: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 of cycle 1 in the absence of disease progression or unacceptable toxicity. Patients then receive fludarabine IV over 30 minutes QD on days 1-5 of cycle 2 and cytarabine IV over 1-3 hours QD on days 1-5 of cycle 2 in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5 of cycle 1 and IMGN632 IV on days 1 and 22 of cycle 1 in the absence of disease progression or unacceptable toxicity. Patients then receive fludarabine IV over 30 minutes QD on days 1-5 of cycle 2, cytarabine IV over 1-3 hours QD on days 1-5 of cycle 2, and IMGN632 IV on days 1 and 22 of cycle 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for the first year, twice a year for year two and yearly visits until five years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients from Children's Oncology Group (COG) sites must be enrolled on APAL2020SC
* Patients must be >= 12 months and less than 22 years of age at the time of study enrollment
* Patient's weight at time of enrollment must be >= 10 kg
* Patients must meet the eligibility in the appropriate Cohort for their diagnosis and disease status

  * Cohort 1 (Phase 1 Monotherapy):

    * Patients must meet all the following criteria:

      * Patient must have bone marrow sample showing >= 5% leukemic blasts by flow cytometry
      * Patient must have been diagnosed with AML, B-ALL, T-ALL, or mixed phenotype acute leukemia (MPAL) meeting one of the following disease criteria:

        * Second or greater relapse OR
        * Disease that is refractory to relapse therapy

          * Refractory to relapse therapy is defined as persistent disease after at least one cycle of induction chemotherapy to treat the relapse disease
      * Patient must have leukemic blasts that are CD123-positive by flow cytometry as determined either by the treating institution or through reference laboratory testing.
  * Cohort 2 (Combination Dose Finding) and Cohort 3 (Randomized Phase 2 Combination):

    * Patients must meet all the following criteria:

      * Patient must have AML in first relapse with a bone marrow sample showing >= 1% leukemic blasts by flow cytometry
      * Patient must have leukemic blasts that are CD123-positive by flow cytometry as determined either by the treating institution or through reference laboratory testing
      * For Cohort 3 only: Patient's AML is not treatment related
  * Central nervous system (CNS) disease - All Cohorts

    * Patients may have status of CNS1, CNS2, CNS3 disease without clinical signs or neurologic symptoms suggestive of CNS leukemia, such as facial nerve palsy, brain/eye involvement or hypothalamic syndrome
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2 (>= 50% Lansky or Karnofsky score). Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. Please refer to the table of myelosuppressive/Anticancer Agents on the COG website: https://www.cogmembers.org/uploadedFiles/Site/Disc/DVL/Documents/TableOfMyelosuppressiveAnti-CancerAgents.pdf. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

  * Cytotoxic chemotherapy: Must not have received within 14 days of entry onto this study, except for hydroxyurea or corticosteroids

    * NOTE: Cytoreduction with hydroxyurea or corticosteroids must be discontinued prior to the start of protocol therapy. Use of steroids for other purposes such as premedication to prevent allergic reaction or during anesthesia is allowed
  * Intrathecal cytotoxic therapy

    * No waiting period is required for patients having received any combination of intrathecal cytarabine, methotrexate, and/or hydrocortisone
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of an antibody-drug conjugate. For unmodified antibodies or T cell engaging antibodies, 2 half-lives must have elapsed before enrollment. Any toxicity related to prior antibody therapy must be recovered to Grade =< 1
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short acting growth factor
  * Radiation therapy (RT):

    * 14 days have elapsed for local palliative RT (small port);
    * >= 84 days must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis;
    * >= 42 days must have elapsed if other substantial bone marrow (BM) radiation
    * For combination therapy arms: Patients must have received =< 13.6 Gy prior radiation to the mediastinum
  * Stem cell infusions:

    * >= 84 days since allogeneic (non-autologous) bone marrow or stem cell transplant (with or without total body irradiation [TBI]) or boost infusion (any stem cell product; not including donor lymphocyte infusion [DLI])
    * No evidence of graft versus host disease (GVHD)
    * Patients must be off medications to treat or prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant for at least 14 days prior to start of protocol treatment
  * Cellular therapy: >= 42 days after the completion of DLI (donor lymphocyte infusion) or any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
* Ejection fraction (EF) of >= 55% or if EF unavailable, shortening fraction (SF) >= 28% by echocardiogram (within 21 days prior to enrollment and start of protocol therapy [repeat if necessary]) AND
* Corrected QTc interval < 500 msec (within 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows (within 7 days prior to enrollment):

  * 1 to < 2 years (age); 0.6 mg/dL (male) 0.6 mg/dL (female)
  * 2 to < 6 years (age); 0.8 mg/dL (male) 0.8 mg/dL (female)
  * 6 to < 10 years (age); 1 mg/dL (male) 1 mg/dL (female)
  * 10 to < 13 years (age); 1.2 mg/dL (male) 1.2 mg/dL (female)
  * 13 to < 16 years (age); 1.5 mg/dL (male) 1.4 mg/dL (female)
  * >= 16 years (age); 1.7 mg/dL (male) 1.4 mg/dL (female)
* Direct bilirubin < 2 mg/dL (< 34 umol/L), (within 7 days prior to enrollment) AND
* Serum glutamate pyruvate transaminase SGPT (alanine aminotransferase [ALT]) =< 135 U/L (within 7 days prior to enrollment)

  * If liver abnormality is due to leukemia infiltrate, the patient will remain eligible

Exclusion Criteria:

* Plans to administer any type of non-protocol prescribed anti-cancer therapy while on protocol directed therapy. For Cohort 1, additional intrathecal therapy is allowed per treating physician's discretion
* Strong inducers or inhibitors of CYP2D6 or CYP3A4 are prohibited for 7 days prior to the 1st dose of IMGN632 to the end of the treatment for both the Phase 1 Monotherapy Dose Finding and pharmacokinetic (PK) and the Combination Dose Finding components of the study. For patients not enrolled in a dose finding portion of the study, concomitant therapy with strong inducers or inhibitors of CYP2D6 or CYP3A4 is STRONGLY discouraged but not prohibited if clinically indicated
* Patients with acute promyelocytic leukemia (APL) or juvenile myelomonocytic leukemia (JMML)
* Patients with Down syndrome
* Patients with isolated extramedullary disease or those with minimal bone marrow disease not meeting the definition of relapsed or relapse refractory as defined above
* Patients with a prior history of Grade 4 VOD/SOS (veno-occlusive disease/sinusoidal obstructive syndrome) or any history of Grade 3 VOD/SOS that, at the discretion of the treating physician, places the patient at unacceptably high risk for future severe VOD/SOS
* Patients who are currently receiving another investigational drug
* Patients receiving medications for treatment of left ventricular systolic dysfunction
* Patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known congenital bone marrow failure syndrome
* Patients with known prior allergy to any of the medications used in protocol therapy
* Patients with documented active, uncontrolled infection at the time of study entry
* Patients with history of Wilson's disease or other copper-related disorder
* Pregnancy and breastfeeding:

  * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
  * Lactating females who plan to breastfeed their infants
  * Sexually active patients of reproductive potential (male and female) who have not agreed to use an effective contraceptive method or abstinence for the duration of their study participation and for 12 weeks after the last dose of IMGN632 or 6 months after last dose of DAUNOrubicin and cytarabine liposome, whichever is longer
* Regulatory requirements

  * All patients and/or their parents or legal guardians must sign a written informed consent
  * All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 12 Months to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of IMGN632 monotherapy (Cohort 1) | During cycle 1 (Each cycle = 42 days)
  Dose limiting toxicities (DLTs) during cycle 1 will be evaluated using a rolling 6 design.
Flow-based overall response rate (ORR) (Cohort 1) | During cycle 1 (Each cycle = 42 days)
  ORR defined as complete remission (CR)/CR with incomplete blood count recovery (CRi)/CR with partial recovery of platelet count (CRp).
RP2D of combination therapy (Cohort 2) | During cycle 1 (Each cycle = 42 days)
  Dose limiting toxicities (DLTs) during cycle 1 combination of DAUNOrubicin and cytarabine liposome and IMGN632 will be evaluated using a rolling 6 design.
Minimal residual disease (MRD) negative flow-based ORR (Cohort 3) | Up to two cycles of IMGN632 with chemotherapy (Each cycle = 42 days)
  Eligible patients will be assessed for MRD negative responses at the end of each cycle of therapy and compared for those receiving therapy including DAUNOrubicin and cytarabine liposome with or without IMGN632. Responders versus non-responders will be classified based on response after up to 2 cycles with a response definition of < 0.01% abnormal blasts by central flow cytometry in a cellular bone marrow. Fisher's Exact test will be used to compare the MRD negative response rate after up to 2 cycles (DAUNOrubicin and cytarabine liposome treatment) followed by fludarabine/cytarabine in pediatric patients with first relapse of acute myeloid leukemia randomized to treatment with or without IMGN632.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the area under the plasma concentration versus time curve (AUC) of IMGN632.
Maximum serum concentration (Cmax) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the maximum serum concentration (Cmax) of IMGN632.
Volume of distribution at steady state (Vss) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the volume of distribution at steady state (Vss) of IMGN632.
Half-life (t1/2) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the half-life (t1/2) of IMGN632.
Clearance (CL) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the clearance (CL) of IMGN632.
Time to reach maximum serum concentration (Tmax) of IMGN632 | Cycles 1 & 2
  Non-compartmental methods will be used to estimate the time to reach maximum serum concentration (Tmax) of IMGN632.

OTHER OUTCOMES:
Morphologic and flow-based CR/CRp/CRi of IMGN632 monotherapy (Cohort 1) | Up to 2 cycles (Each cycle = 42 days)
  Patients enrolled onto the monotherapy Phase 1 arm will be grouped by disease type (acute myeloid leukemia [AML], B-cell acute lymphoblastic leukemia [ALL], early thymic precursor [ETP] T-cell ALL and mixed phenotype acute leukemia [MPAL]) and the anti-leukemic activity of IMGN632 monotherapy will be described.
Rates of MRD negative response of IMGN632 monotherapy (Cohort 1) | Up to 2 cycles (Each cycle = 42 days)
  Patients enrolled onto the monotherapy Phase 1 arm will be grouped by disease type (AML, B-cell ALL, ETP T-cell ALL and MPAL) and the anti-leukemic activity of IMGN632 monotherapy will be described.
Event-free survival (EFS) of IMGN632 monotherapy (Cohort 1) | Up to 5 years
  Patients enrolled onto the monotherapy Phase 1 arm will be grouped by disease type (AML, B-cell ALL, ETP T-cell ALL and MPAL) and the anti-leukemic activity of IMGN632 monotherapy will be described.
Overall survival (OS) of IMGN632 monotherapy (Cohort 1) | Up to 5 years
  Patients enrolled onto the monotherapy Phase 1 arm will be grouped by disease type (AML, B-cell ALL, ETP T-cell ALL and MPAL) and the anti-leukemic activity of IMGN632 monotherapy will be described.
EFS for patients with first relapse of AML (Cohort 3) | Up to 5 years
OS for patients with first relapse of AML (Cohort 3) | Up to 5 years
Cumulative incidence of relapse for patients with first relapse of AML (Cohort 3) | Up to 5 years
Use of stem cell transplant after protocol therapy (Cohort 3) | Up to 5 years
  Will be collected and the rate of subsequent stem cell transplant will be described by treatment arm. This will include data regarding the conditioning regimen used, stem cell donor source and transplant related toxicities such as veno-occlusive disease.
Incidence of adverse events (Cohort 3) | Up to 5 years
  Will be summarized by treatment arm for patients with first relapse of AML treated during the randomized Phase 2.
CD123 expression | Up to 5 years
  CD123 expression on leukemic blasts will be analyzed at Hematologics, Inc. (Seattle, Washington [WA]) by multi-dimensional flow cytometry (MDF) utilizing a "difference from normal" flow cytometric technique. CD123 mean fluorescent intensity (MFI) will be quantified and converted to molecules per cell (MPC) using CD4 MFI on T cells as a reference. CD123 MPC will be assessed on bone marrow (or peripheral blood samples if bone marrow not available) at initial diagnosis and after cycle 1 of treatment for patients with first relapse of AML treated on the randomized phase 2 portion of this study. Outcomes, including OS, EFS, and MRD negative CR after cycle 1, will be correlated with CD123 MPC and compared between the groups of patients who did and did not receive the investigational therapy IMGN632 using Cox and logistic regression models.
Cumulative incidence of left ventricular systolic dysfunction (LVSD) | Up to 1 year post AML relapse
  Will be estimated with subsequent relapse and death considered competing events. Cox regression will be used to estimate adjusted hazard ratio (HR) comparing EFS and OS in patients with LVSD relative to patients with no LVSD. LVSD will be treated as a time-varying exposure introduced on the first occurrence during/ following salvage therapy. HRs will be determined separately for infection-associated or not infection-associated events. Exploratory analyses will be performed to assess the differential impact of infection vs. non-infection associated LVSD on survival.
Incidence of adverse events (All Cohorts) | Up to 5 years
  Will be described by summarizing adverse events reported for patients on protocol therapy. Long-term safety will include assessment and summary of the following: all toxicities reported (including any death that can be attributed possibly, probably, or definitely to protocol therapy and is not due to cancer recurrence and any secondary malignancy that can be attributed possibly, probably, or definitely to protocol therapy), all Grade 5 events regardless of attribution, all grades of sinusoidal obstructive syndrome (SOS)/veno-occlusive disease (VOD) and Grade 3 or greater of the cardiac toxicities ventricular arrhythmia and left ventricular systolic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Kutny, Principal Investigator — Children's Oncology Group